CLINICAL TRIAL: NCT00710801
Title: Randomized, Open-label Study to Evaluate the Hepatitis C Virus (HCV) Burden in Patients Receiving Cyclosporine (Neoral or CSA) Versus Tacrolimus (Prograf) in de Novo Liver Recipients Receiving Mycophenolate Sodium (Myfortic): Assessment of Biomarkers for Recurrent HCV Infection Post-liver Transplantation
Brief Title: Assessment of Biomarkers for Recurrent HCV Infection Post-liver Transplantation
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: COLO400A2427
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Virus; HCV; Liver Transplant; Cyclosporine; Tacrolimus; Myfortic
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Tissue

SUMMARY:
The purpose of this study is to learn about how different immunosuppressant therapies impact on recurrent hepatitis C virus infection in the new liver after liver transplant. We will be evaluating if Cyclosporin A has a superior effect against recurrent Hepatitis C virus (HCV) infection than Tacrolimus.

DETAILED DESCRIPTION:
We will address the hypothesis that CSA has a superior antiviral effect against HCV than Tacrolimus by assessing serial HCV RNA levels in serum. We plan to address the hypothesis that CSA is more efficient in limiting viremia than Tacrolimus and that viremia is predictive of long-term clinical outcome of hepatic fibrosis that is known to impact on both graft and patient survival

ELIGIBILITY:
Inclusion Criteria:

* About to undergo a primary liver transplant (including living donor, split liver) and are HCV positive.
* Willing and capable of giving written consent for study participation
* Expected to be capable of study participation for full 24 months post-transplantation.
* Allograft biopsies will be possible
* Expected use of calcineurin inhibitor (Neoral or Tacrolimus) as primary immunosuppression An immunosuppressive regimen consisting of a calcineurin inhibitor (Neoral or Tacrolimus) in combination with Simulect and MYCOPHENOLATE SODIUM

Exclusion Criteria:

* This is a multi-organ transplant or if the patient has previously been transplanted with any other organ.
* This is a liver transplant from a non-heart beating donor.
* This is an ABO incompatible transplant.
* Patients with serum creatinine level > 250 umol/L.
* The recipient is seropositive for human immunodeficiency virus (HIV) antibodies.
* Fulminant liver failure is the reason for transplant.
* Patient is participating in other clinical trial involving exploratory drug
* There is a known malignancy, or a history of malignancy, other than successfully treated non-metastatic basal or squamous cell carcinoma of the skin, or hepatocellular carcinoma less than 5 cm meeting Milan criteria for transplantation5.
* The patient is being transplanted for hepatic malignancy with greater than 5 known lesions.
* Severe coexisting disease is present or if any unstable medical condition is present which could affect the study objectives.
* A female transplant candidate is pregnant, lactating or of childbearing potential and not practicing an acceptable method of contraception.
* An unlicensed drug or therapy has been administered within one month prior to study entry or if such therapy is to be instituted post-transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV positive patients undergoing orthotopic liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L Mason, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada